CLINICAL TRIAL: NCT02279771
Title: Multicenter Randomized Controlled Trial of Transanal Reinforcement of Low Rectal Anastomosis Versus Protective Ileostomy in the Prevention of Anastomotic Leak After Rectal Cancer Surgery
Brief Title: Transanal Reinforcement of Low Rectal Anastomosis in Rectal Cancer Surgery
Acronym: LessStoReS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Donato F Altomare (Network)
Responsible Party: Sponsor-Investigator, Donato F Altomare, Associate professor, Societa Italiana di Chirurgia ColoRettale
Organization: Societa Italiana di Chirurgia ColoRettale (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Siccr/2014
Record Dates: First submitted 2014-10-29; First posted 2014-10-31 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Rectal Cancer
Keywords: colorectal anastomosis; anastomotic leak; ileostomy; complications
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- transanal anastomotic reinforcement (Active Comparator): Low anterior resection with TME plus anastomotic transanal reinforcement without protective ileostomy/colostomy (transanal anastomotic reinforced arm:TAR-LAR)
  Interventions: Procedure: transanal anastomotic reinforcement; Device: a circular anal dilator (CAD)
- protective ileostomy group (Active Comparator): Standard low anterior resection with TME plus protective ileostomy/colostomy (S-LAR)
  Interventions: Procedure: protective ileostomy group

INTERVENTIONS:
Procedure: transanal anastomotic reinforcement — a circular anal dilator (CAD) of 34mm in diameter will be introduced into the anus to facilitate the transanal introduction of the 29-31 circular stapler. The stapler shaft will be introduced trying to avoid the stapler line and connected with the anvil of the prepared proximal colon and then fired.
  Patients selected on the TAR-LAR arm will have the stapled suture reinforced by 6 supplemental full thickness stitches in vycril 3/0 placed transanally with the aid of a semicircular valve introduced into the CAD (Epo Flier, SapiMed SPA, Alessandria, Italy), at hours 2-4-6-8-10-12.
  Arms: transanal anastomotic reinforcement
Procedure: protective ileostomy group — S-LAR patients will had a standard lateral protective ileostomy in the right iliac region or a colostomy in the left region.
  Arms: protective ileostomy group
Device: a circular anal dilator (CAD) — Epo Flier, SapiMed SPA, Alessandria, Italy
  Arms: transanal anastomotic reinforcement

SUMMARY:
Anastomotic leak after low rectal cancer surgery occurs between 3 and 24% of the cases and is a severe complication leading to sepsis, permanent colostomy, higher risk of local cancer recurrence and eventually death. In order to prevent this complication a protecting diverting stoma is usually fashioned with consequent morbidity due to the stoma and its closure and severe impact on patients' quality of life. This prospective, multi-center, parallel-arm, randomized controlled equivalence trial is aimed to demonstrate whether a transanal reinforcement of the suture line can prevent anastomotic leakage after low rectal cancer surgery thus avoiding the need for a covering ileostomy

ELIGIBILITY:
Inclusion Criteria:

* Resectable, histologically proven primary adenocarcinoma of the medium-low rectum without internal and/or external sphincter muscle involvement.

Distal margin of the tumor at least 6 cm form the anal verge

Staged as follows prior to neoadjuvant chemoradiation:

Stage T2 - T4 at MRI N0-2 at MRI M0/M1 at CT scan Patient classified T3-T4 must undergo neoadjuvant chemoradiation with at least 8 weeks delay of surgery

Exclusion Criteria:

* Squamous cell carcinoma
* Adenocarcinoma Stage T1,
* T4 with one of the following:

with pelvic side wall involvement requiring sacrectomy requiring prostatectomy (partial or total)

* Unresectable primary rectal cancer or Inability to complete R0 resection.
* Rectal cancer under 6 cm from the anal verge requiring colo-anal anastomosis
* Recurrent rectal cancer
* Previous pelvic malignancy
* Inability to sign informed consent
* Pregnancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-01; Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
anastomotic leak | 30 postoperative days
  anastomoltic leak will be checked by barium enema after 30 days from the low rectal anastomosis

SECONDARY OUTCOMES:
duration of the two operations | Intraoperative
  the duration in minutes of the two types of operation
Number of overall postoperative complications | 30 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Arcangelo Picciariello, MD, Principal Investigator — Societa Italiana di Chirurgia ColoRettale
Locations (1):
- Bari, Italy

REFERENCES:
- [Background] Cong ZJ, Hu LH, Bian ZQ, Ye GY, Yu MH, Gao YH, Li ZS, Yu ED, Zhong M. Systematic review of anastomotic leakage rate according to an international grading system following anterior resection for rectal cancer. PLoS One. 2013 Sep 25;8(9):e75519. doi: 10.1371/journal.pone.0075519. eCollection 2013. PMID 24086552
- [Background] Siegel R, Naishadham D, Jemal A. Cancer statistics, 2013. CA Cancer J Clin. 2013 Jan;63(1):11-30. doi: 10.3322/caac.21166. Epub 2013 Jan 17. PMID 23335087
- [Background] Heald RJ, Husband EM, Ryall RD. The mesorectum in rectal cancer surgery--the clue to pelvic recurrence? Br J Surg. 1982 Oct;69(10):613-6. doi: 10.1002/bjs.1800691019. PMID 6751457
- [Background] Karanjia ND, Corder AP, Bearn P, Heald RJ. Leakage from stapled low anastomosis after total mesorectal excision for carcinoma of the rectum. Br J Surg. 1994 Aug;81(8):1224-6. doi: 10.1002/bjs.1800810850. PMID 7953369
- [Background] Fazio VW, Zutshi M, Remzi FH, Parc Y, Ruppert R, Furst A, Celebrezze J Jr, Galanduik S, Orangio G, Hyman N, Bokey L, Tiret E, Kirchdorfer B, Medich D, Tietze M, Hull T, Hammel J. A randomized multicenter trial to compare long-term functional outcome, quality of life, and complications of surgical procedures for low rectal cancers. Ann Surg. 2007 Sep;246(3):481-8; discussion 488-90. doi: 10.1097/SLA.0b013e3181485617. PMID 17717452
- [Background] Matthiessen P, Hallbook O, Andersson M, Rutegard J, Sjodahl R. Risk factors for anastomotic leakage after anterior resection of the rectum. Colorectal Dis. 2004 Nov;6(6):462-9. doi: 10.1111/j.1463-1318.2004.00657.x. PMID 15521937
- [Background] Gong JP, Yang L, Huang XE, Sun BC, Zhou JN, Yu DS, Zhou X, Li DZ, Guan X, Wang DF. Outcomes based on risk assessment of anastomotic leakage after rectal cancer surgery. Asian Pac J Cancer Prev. 2014;15(2):707-12. doi: 10.7314/apjcp.2014.15.2.707. PMID 24568483
- [Background] Rullier E, Laurent C, Garrelon JL, Michel P, Saric J, Parneix M. Risk factors for anastomotic leakage after resection of rectal cancer. Br J Surg. 1998 Mar;85(3):355-8. doi: 10.1046/j.1365-2168.1998.00615.x. PMID 9529492
- [Background] Mirnezami A, Mirnezami R, Chandrakumaran K, Sasapu K, Sagar P, Finan P. Increased local recurrence and reduced survival from colorectal cancer following anastomotic leak: systematic review and meta-analysis. Ann Surg. 2011 May;253(5):890-9. doi: 10.1097/SLA.0b013e3182128929. PMID 21394013
- [Background] Branagan G, Finnis D; Wessex Colorectal Cancer Audit Working Group. Prognosis after anastomotic leakage in colorectal surgery. Dis Colon Rectum. 2005 May;48(5):1021-6. doi: 10.1007/s10350-004-0869-4. PMID 15789125
- [Background] Testini M, Gurrado A, Portincasa P, Scacco S, Marzullo A, Piccinni G, Lissidini G, Greco L, De Salvia MA, Bonfrate L, Debellis L, Sardaro N, Staffieri F, Carratu MR, Crovace A. Bovine pericardium patch wrapping intestinal anastomosis improves healing process and prevents leakage in a pig model. PLoS One. 2014 Jan 29;9(1):e86627. doi: 10.1371/journal.pone.0086627. eCollection 2014. PMID 24489752
- [Background] Baek SJ, Kim J, Kwak J, Kim SH. Can trans-anal reinforcing sutures after double stapling in lower anterior resection reduce the need for a temporary diverting ostomy? World J Gastroenterol. 2013 Aug 28;19(32):5309-13. doi: 10.3748/wjg.v19.i32.5309. PMID 23983434
- [Background] Senagore A, Lane FR, Lee E, Wexner S, Dujovny N, Sklow B, Rider P, Bonello J; Bioabsorbable Staple Line Reinforcement Study Group. Bioabsorbable staple line reinforcement in restorative proctectomy and anterior resection: a randomized study. Dis Colon Rectum. 2014 Mar;57(3):324-30. doi: 10.1097/DCR.0000000000000065. PMID 24509454
- [Background] Gastinger I, Marusch F, Steinert R, Wolff S, Koeckerling F, Lippert H; Working Group 'Colon/Rectum Carcinoma'. Protective defunctioning stoma in low anterior resection for rectal carcinoma. Br J Surg. 2005 Sep;92(9):1137-42. doi: 10.1002/bjs.5045. PMID 15997447
- [Background] Matthiessen P, Hallbook O, Rutegard J, Simert G, Sjodahl R. Defunctioning stoma reduces symptomatic anastomotic leakage after low anterior resection of the rectum for cancer: a randomized multicenter trial. Ann Surg. 2007 Aug;246(2):207-14. doi: 10.1097/SLA.0b013e3180603024. PMID 17667498
- [Background] Bafford AC, Irani JL. Management and complications of stomas. Surg Clin North Am. 2013 Feb;93(1):145-66. doi: 10.1016/j.suc.2012.09.015. PMID 23177069
- [Background] Chow A, Tilney HS, Paraskeva P, Jeyarajah S, Zacharakis E, Purkayastha S. The morbidity surrounding reversal of defunctioning ileostomies: a systematic review of 48 studies including 6,107 cases. Int J Colorectal Dis. 2009 Jun;24(6):711-23. doi: 10.1007/s00384-009-0660-z. Epub 2009 Feb 17. PMID 19221766
- [Background] Perez Dominguez L, Garcia Martinez MT, Caceres Alvarado N, Toscano Novella A, Higuero Grosso AP, Casal Nunez JE. Morbidity and mortality of temporary diverting ileostomies in rectal cancer surgery. Cir Esp. 2014 Nov;92(9):604-8. doi: 10.1016/j.ciresp.2013.12.011. Epub 2014 Jun 23. English, Spanish. PMID 24969349
- [Background] Altomare DF, Pannarale OC, Lupo L, Palasciano N, Memeo V, Rubino M. Protective colostomy closure: the hazards of a "minor" operation. Int J Colorectal Dis. 1990 May;5(2):73-8. doi: 10.1007/BF00298472. PMID 2358740
- [Background] Chiu A, Chan HT, Brown CJ, Raval MJ, Phang PT. Failing to reverse a diverting stoma after lower anterior resection of rectal cancer. Am J Surg. 2014 May;207(5):708-11; discussion 711. doi: 10.1016/j.amjsurg.2013.12.016. Epub 2014 Mar 12. PMID 24791631
- [Derived] Altomare DF, Delrio P, Shelgyn Y, Rybakov E, Vincenti L, De Fazio M, Simone M, Graziano G, Picciariello A. Transanal reinforcement of low rectal anastomosis versus protective ileostomy after total mesorectal excision for rectal cancer. Preliminary results of a randomized clinical trial. Colorectal Dis. 2021 Jul;23(7):1814-1823. doi: 10.1111/codi.15685. Epub 2021 May 10. PMID 33891798